CLINICAL TRIAL: NCT02390791
Title: Developing New Technologies to Improve ADHD Medication Continuity
Brief Title: New Technologies to Help Manage ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R34MH101155 (NIH); R34MH101155 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-18 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- enhanced myADHDportal.com (Experimental): Version of the myADHDportal.com web software enhanced with family-management support to enable parents to be active partners in optimizing and maintaining medication continuity for their child
  Interventions: Other: enhanced myADHDportal.com
- treatment as usual standard portal (Active Comparator): Standard version of myADHDportal.com web software
  Interventions: Other: treatment as usual standard portal

INTERVENTIONS:
Other: enhanced myADHDportal.com — Version of the myADHDportal.com web software enhanced with family-management support to enable parents to be active partners in optimizing and maintaining medication continuity for their child
  Arms: enhanced myADHDportal.com
Other: treatment as usual standard portal — Standard version of myADHDportal.com web software
  Arms: treatment as usual standard portal

SUMMARY:
Cluster randomized controlled trial to evaluate the general effectiveness of intervention compared to control on medication continuity as measured by prescriptions written and other more proximal outcomes during the first six months of treatment.

DETAILED DESCRIPTION:
This cluster randomized controlled trial will evaluate the general effectiveness of the intervention (e.g. enhanced myADHDportal.com), compared to control (e.g. treatment as usual standard portal), on medication continuity as measured by prescriptions written and other more proximal outcomes during the first six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children are eligible to participate if

  1. their child receives ADHD care at one of the pediatric primary care practices that is partnering to conduct this trial
  2. child being registered on myADHDportal.com to initiate child assessment of ADHD
  3. child age 6-10 years
  4. child must not have been previously treated with ADHD medication
  5. child prescribed ADHD medication within 12 months of enrolling in the study

Exclusion Criteria:

* Unable to read and speak English

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, MEd, MSc, Principal Investigator — Cincinnati Children's
Locations (1):
- William B Brinkman, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Started | 40 | 45
Completed | 40 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal | Total
Number analyzed (Participants) | 40 | 45 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.88 (1.34) | 7.96 (1.23) | 7.92 (1.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 28 | 34 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 37 | 39 | 76
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 6 | 13
  White | 30 | 33 | 63
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Medication Continuity: The Number of Days Covered With Medicine
Description: the number of days covered with medicine will be calculated from audit of prescriptions written
Time Frame: first 6 months of treatment
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 40 | 45
Days | 108.8 (45.8) | 133.3 (50.9)
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.04, generalized linear model; assuming a Poisson distribution with a log link function

2. Secondary Outcome: Parent-reported Necessity to Concerns Differential (Beliefs About Medication Scale)
Description: Necessity to concerns differential score, range -4 to 4, positive scores mean necessity outweighs concerns, negative scores mean that concerns outweigh beliefs about necessity
Time Frame: 6 months after starting treatment
Population: population who completed this outcome assessment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 23 | 24
score on a scale | 0.44 [-1.18 to 1.11] | -0.06 [-0.52 to 0.86]
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Parent-reported Decisional Conflict (Decisional Conflict Scale)
Description: Total score calculated from parent-report on the Decisional Conflict Scale, range 0 to 100; higher scores are worse
Time Frame: 6 months after starting treatment
Population: population who completed this outcome assessment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 23 | 25
score on a scale | 14.06 [6.25 to 29.69] | 20.31 [14.06 to 26.56]
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Parent Trust in Provider (Trust in Provider Scale)
Description: Total score calculated from parent-report on the Trust in Provider Scale, range 10 to 50 with higher scores better (more trust)
Time Frame: 6 months after starting treatment
Population: population who completed this outcome assessment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 23 | 24
score on a scale | 45.0 [38.0 to 48.0] | 41.5 [39.0 to 46.5]
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Working Alliance Inventory
Description: range 12-60, higher scores better (more alliance)
Time Frame: 6 months after starting treatment
Population: population who completed this outcome assessment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 23 | 24
score on a scale | 50.0 [44.0 to 55.0] | 46.0 [44.0 to 49.5]
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Parent Perceived Social Support (Perceived Social Support Scale)
Description: Total score calculated from parent-report on the Perceived Social Support Scale, range 12-84, higher score better (more social support)
Time Frame: 6 months after starting treatment
Population: population who completed this outcome assessment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 23 | 24
score on a scale | 54.00 [42.0 to 72.0] | 68.95 [44.0 to 72.0]
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Parent Distress (Parenting Stress Index - Short Form)
Description: Parental distress subscale score calculated from the Parenting Stress Index - Short Form; range 36-180, higher scores is worse (more stress)
Time Frame: 6 months after starting treatment
Population: population who completed this outcome assessment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 22 | 23
score on a scale | 75.57 [55.0 to 92.0] | 74.00 [56.0 to 93.0]
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Participants With Side Effects Rated by Parents as Moderate or Severe on the Pittsburgh Side Effects Rating Scale
Description: Number of Participants with side effects rated by parents as moderate or severe on the Pittsburgh Side Effects Rating Scale
Time Frame: 6 months after starting treatment
Population: population who completed this outcome assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 23 | 25
Participants | 13 | 9
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.15, Chi-squared

9. Secondary Outcome: Total Number of myADHDportal.Com Log-ins by Parent
Time Frame: 6 months after starting treatment
Measure: Mean (Standard Deviation); unit: logins
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 40 | 45
logins | 11.33 (13.84) | 8.47 (7.53)
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.48, generalized linear model

10. Secondary Outcome: Total Number of Measures Completed by Parents to Track Child Response to Treatment
Time Frame: 6 months after starting treatment
Measure: Mean (Standard Deviation); unit: measures
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
Number analyzed (Participants) | 40 | 45
measures | 2.50 (3.37) | 2.31 (3.00)
Statistical Analysis 1: Comparison: Enhanced myADHDportal.Com vs Treatment as Usual Standard Portal; Test type: Superiority; p = 0.71, generalized linear model

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Enhanced myADHDportal.Com | Treatment as Usual Standard Portal
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/45
Other Adverse Events (participants affected / at risk) | 0/40 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02390791/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02390791/SAP_001.pdf